CLINICAL TRIAL: NCT07009444
Title: The Role of Mental Imagery on Approach Motivation and Behavioral Engagement in Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Christoph Benke, Principal Investigator, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DARE
Record Dates: First submitted 2025-05-14; First posted 2025-06-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Social Anxiety; Social Phobia
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation + Prospective Mental-Imagery Task (Experimental): Prospective mental imagery of post-exposure experience
  Interventions: Behavioral: Psychoeducation; Behavioral: Prospective Mental Imagery
- Psychoeducation (Active Comparator)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Psychoeducation — Providing information about social anxiety, role of safety and avoidance behaviors in maintaining social anxiety, rationale for exposure to feared social situations
Behavioral: Prospective Mental Imagery — A standard imagination script is recounted in which participants have successfully mastered the socially feared situation
  Arms: Psychoeducation + Prospective Mental-Imagery Task

SUMMARY:
Efficacy of an online intervention aimed at enhancing both approach motivation and behavioral engagement in facing anxiety-provoking social situations among individuals with heightened social anxiety is investigated. Upon receiving psychoeducation, participants will either undergo a prospective mental-imagery task or no additional task. The intervention's efficacy will be assessed by ratings of experienced and expected pleasure, approach motivation as well as self-reported engagement with feared situation one week later.

DETAILED DESCRIPTION:
Although exposure therapy is widely considered the gold standard for treating anxiety disorders, its effectiveness is often hindered by treatment discontinuation. Many individuals avoid facing feared situations, yet exposure is crucial for successful extinction learning. Therefore, there is a need for strategies to enhance both approach motivation and behavioral engagement in anxiety-provoking situations. Within the depression literature, imagery-based interventions have already gained some support in increasing motivation and behavioral engagement in pleasurable activities through enhancement of reward anticipation as well as anticipatory and anticipated pleasure ('motivational amplifier' hypothesis). Considering that social anxiety is characterized by disruptions in motivational and reward processes, prospective mental imagery may strengthen approach motivation and behavioral engagement in exposure to socially feared situations. Thus, the present online study will investigate the effect of a prospective mental-imagery task on approach motivation and behavioral engagement in socially anxious individuals. Following psychoeducation, participants in the experimental group will vividly imagine having successfully mastered the fear-provoking situation. The control group will receive only psychoeducation. Approach motivation as well as reward anticipation, anticipated and anticipatory pleasure will be assessed before and after the psychoeducation and imagery task. Engagement with the feared social situation will be assessed one week later. The aim of this randomized controlled trial in healthy individuals with heightened social anxiety is to investigate whether prospective mental imagery is effective in enhancing self-reported motivation and engagement with feared situation compared to a psychoeducation-only control group. In an exploratory analysis, we will investigate whether individuals' levels of reward sensitivity and anhedonia influence the effectiveness of prospective imagery training.

ELIGIBILITY:
Inclusion Criteria:

* Elevated score on Mini-Social Phobia Inventory (Mini-SPIN) > 6

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Anticipatory Pleasure | Baseline (prior to the assigned intervention) and immediately post-intervention (following prospective mental imagery or psychoeducation)
  2-item questionnaire on a scale 0 (not at all) to 100 (extremely) assessing current pleasure when imaging approaching and having approached the feared situation.
Anticipated Pleasure | Baseline (prior to the assigned intervention) and immediately post-intervention (following prospective mental imagery or psychoeducation)
  2-item questionnaire on a scale 0 (not at all) to 100 (extremely) assessing expected pleasure when approaching and having approached the feared situation.
Reward Anticipation | Baseline (prior to the assigned intervention) and immediately post-intervention (following prospective mental imagery or psychoeducation)
  2-item questionnaire on a scale 0 (not at all) to 100 (extremely) assessing expected reward related to approaching and having approached the feared situation.
Motivation | Baseline (prior to the assigned intervention) and immediately post-intervention (following prospective mental imagery or psychoeducation)
  Self-reported motivation to approach the feared situation on a scale of 0 (not at all) to 100 (extremely).
Frequency of Exposure | Post-treatment (i.e., 7 days after baseline)
  Self-reported frequency of exposure to the feared situation. Scale: 0 to 10, indicating the frequency of exposure to the feared situation.

SECONDARY OUTCOMES:
Social Phobia Inventory (SPIN) | Change from baseline to post-treatment (i.e., 7 days)
  17-item questionnaire on a 5-point Likert scale (0 = 'not at all'; 4 = 'extremely') assessing symptom severity related to social anxiety (i.e., fear, avoidance, physical symptoms). Total range score: 0 to 68. Higher scores indicating greater severity of social anxiety.
Liebowitz Social Anxiety Scale (LSAS) | Change from baseline to post-treatment (i.e., 7 days)
  24-item questionnaire on a 4-point Likert scale (fear: 0 = 'none'; 3 = 'severe'; avoidance: 0 = 'never'; 3 = 'usually') assessing both fear/anxiety and avoidance of social situations, respectively. Total range score: 0 to 144. Higher scores indicating greater fear and avoidance as well as severity of social anxiety.
Patient Health Questionnaire-9 (PHQ-9) | Change from baseline to post-treatment (i.e., 7 days)
  9-item questionnaire on a 4-point Likert scale (0 = 'not at all'; 3 = 'nearly every day') assessing the presence and severity of depressive symptoms. Total range score: 0 to 27. Higher scores indicating more severe depression.
Positive and Negative Affect Schedule (PANAS) | Change from baseline to post-treatment (i.e., 7 days)
  20-item questionnaire on a 5-point Likert scale (0 = 'not at all'; 4 = 'extremely') assessing the presence and intensity of both positive and negative emotions. Total score range for positive affect (PA) and negative affect (NA), respectively: 0 to 50. Higher scores indicate on either scale indicate a higher level of that emotion.
BIS/BAS Scales | Baseline
  24-item questionnaire on a 4-point Likert scale (1 = 'strongly disagree'; 4 = 'strongly agree') assessing an individual's tendency toward reward-seeking and punishment-avoidance behavior. Total score range BIS: 7 to 25. Higher scores indicating an increased sensitivity to threats or punishment (BIS). Total score range BAS: 13 to 52. Higher scores indicating a greater propensity to seek rewards and engage in approach behavior.
Temporal Experience of Pleasure Scale (TEPS) | Baseline
  18-item questionnaire on a 6-point Likert scale (1 = 'strongly disagree'; 6 = 'strongly agree') assessing anticipatory and consummatory pleasure. Total score range: 18 to 108. Higher total scores indicating a greater capacity for pleasure.
Vividness of Mental Imagination | Immediately after prospective mental imagery at baseline
  Vividness of imagination on a scale from 0 (not at all) to 100 (extremely vivid) assessed immediately after imagination exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Germany Philipps University, Marburg, Germany

REFERENCES:
- [Background] Hallford DJ, Farrell H, Lynch E. Increasing anticipated and anticipatory pleasure through episodic thinking. Emotion. 2022 Jun;22(4):690-700. doi: 10.1037/emo0000765. Epub 2020 Jun 18. PMID 32551746
- [Background] Renner F, Werthmann J, Paetsch A, Bar HE, Heise M, Bruijniks SJE. Prospective Mental Imagery in Depression: Impact on Reward Processing and Reward-Motivated Behaviour. Clin Psychol Eur. 2021 Jun 18;3(2):e3013. doi: 10.32872/cpe.3013. eCollection 2021 Jun. PMID 36397959
- [Background] Renner F, Murphy FC, Ji JL, Manly T, Holmes EA. Mental imagery as a "motivational amplifier" to promote activities. Behav Res Ther. 2019 Mar;114:51-59. doi: 10.1016/j.brat.2019.02.002. Epub 2019 Feb 5. PMID 30797989
- [Background] Ji JL, Geiles D, Saulsman LM. Mental imagery-based episodic simulation amplifies motivation and behavioural engagement in planned reward activities. Behav Res Ther. 2021 Oct;145:103947. doi: 10.1016/j.brat.2021.103947. Epub 2021 Aug 15. PMID 34433114